CLINICAL TRIAL: NCT05140460
Title: Cultural Pride Reinforcement for Early School Readiness: A Quasi-Experimental Trial
Brief Title: Cultural Pride Reinforcement for Early School Readiness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Ashaunta Anderson, Assistant Professor of Pediatrics, Children's Hospital Los Angeles
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HS-17-139
Record Dates: First submitted 2021-11-08; First posted 2021-12-01 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: School Readiness; Racial Socialization; Child Development
Keywords: Racial Socialization; Ethnic Socialization; Early Childhood; Literacy; Child Development
MeSH Terms: conditions — Literacy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Behavioral: Cultural Pride Reinforcement for Early School Readiness (CPR4ESR)
- Control (Active Comparator)
  Interventions: Behavioral: Reach Out and Read (ROR)

INTERVENTIONS:
Behavioral: Cultural Pride Reinforcement for Early School Readiness (CPR4ESR) — The intervention entails distribution of a children's book with a cultural pride theme and the cultural pride parent book-sharing guide. Intervention participants select and receive a developmentally appropriate (baby, toddler, or preschool) book that features African American, Latino, Asian or diverse cultural pride perspectives.
  Arms: Intervention
Behavioral: Reach Out and Read (ROR) — The control condition involves distribution of a standard ROR book and book-sharing advice. Distributed books are developmentally appropriate (baby, toddler, or preschool).
  Arms: Control

SUMMARY:
Minority children disproportionately experience racial bias, which is linked to school failure, toxic stress, and health disparities. In contrast, a type of racial socialization called cultural pride reinforcement has been associated with positive academic, behavioral, and mental health outcomes. A clinic-based intervention to boost cultural pride may help parents foster resilience in their young children against the negative effects of racial bias. The investigators evaluated the extent to which a standard clinic-based early literacy program (Reach Out and Read (ROR)) and a similar program enhanced with cultural pride content (Cultural Pride Reinforcement for Early School Readiness (CPR4ESR)) are associated with improved cultural pride reinforcement practices, child development, family-provider communication, and health care utilization. Given the high representation of young children of color in the sample, the investigators hypothesized better outcomes among those who received the culturally tailored CPR4ESR program compared to those who received the standard ROR program.

DETAILED DESCRIPTION:
In order to evaluate parental delivery of cultural pride messages, child development, and health services outcomes, 106 parents of children ages 6 months to 5 years old were recruited from two child-serving health institutions in Southern California. This study utilized both an intervention group (n=67) and a control group (n=39). Recruitment and baseline intervention for this study took place on the same day, with one 3-month follow-up conducted over the telephone, and a 1-year post-enrollment review of the child's medical chart. Only a subset (n=14) participated in the medical chart review. Details of the study methodology are provided below.

Recruitment Parents were recruited from two child-serving community health clinics in Southern California. Participants were at least 18 years of age, had a child who was between 6 months and 5 years of age, was of African American, Asian, Latino race/ethnicity or diverse cultural perspective, and reported a primary language that was English or Spanish. Potential participants were identified by the health clinics' coordinating research staff and the clinical pediatrics team. Research assistants (RAs) from the study conferred with the medical staff for each pediatric team to review participant eligibility. The pediatric team distributed the study flyer to those parents who met study eligibility at their scheduled well-child or sick-child visit. Additionally, study flyers were posted at the clinic. Recruitment script and informed consent took approximately 10 minutes.

Intervention Treatment Assignment Participants comprising the intervention group and the control group were determined by designating all participating parents with office visits on even days of the month to the intervention group and all participating parents with office visits on odd days of the month to the control group.

Intervention Group The intervention entails distribution of a children's book with a cultural pride theme, the cultural pride parent book-sharing guide, and the study survey. Consented intervention participants selected and received a developmentally appropriate (baby, toddler, or preschool) book from the RA that featured African American, Latino, Asian, or diverse cultural pride perspectives. All books selected for distribution in the intervention group were vetted through a community advisory board. The cultural pride books differ from the standard ROR books distributed at office visits in that the ROR books address age-related developmental and interactive content, but do not focus on or require specific images and narratives reflective of racial, ethnic, or cultural perspectives in their content. Participating parents were asked to complete the study survey. The survey collected information on demographics, racial socialization (including cultural pride reinforcement), child development, and family-provider communication. Portions of the survey used a 5-point Likert scale to rate the extent to which parents agreed or disagreed with each item. The survey was administered via paper and pencil during the initial intervention in the clinic-designated research room. The RA remained in the room with the participants to address any questions participants may have had when completing the survey. The survey was translated into Spanish. The intervention took approximately 30 minutes: 10 minutes for recruitment/study information and consent, and 20 minutes for book material distribution and review, and survey. Confidentiality of data collected for the survey was maintained through the use of codes.

Control Group The control condition involves distribution of standard ROR book and book-sharing advice, and the study survey. Consented participants received the standard ROR reading advice and a ROR book. Some books from the standard ROR book list may include images reflective of study participants, but without a direct cultural pride message; therefore, books selected from the ROR children's book list for this study were reviewed and selected by the study PI in order to exclude any ROR books for distribution that may resemble cultural pride books. The comparison group was asked to complete the same study survey as the intervention group using the protocol described above.

Three Month Follow-Up Survey Three months following the initial intervention date at clinics with the intervention and control group participants, RAs conducted follow-up telephone calls to participants. Participants were asked, via phone, to complete the same survey as before with 1 additional question to assess feedback on the study experience. For the follow-up survey, participants were read the questions over the phone (in English or Spanish) and their responses documented on a paper survey by RAs. Confidentiality of data collected for the survey was maintained through the use of codes. The follow-up survey took approximately 10 minutes to complete.

One-Year Chart Review In the year following enrollment, clinic personnel reviewed the medical charts of the children whose parents participated in the study and agreed to the optional chart review. Chart reviews identified subsequent records for: number and type of well-child and sick-child visits, dates of office visits, vaccines status at the 1-year mark, and if documented, follow-up visits and diagnosis from emergency room care. During the initial recruitment and intervention at the office visit those participating consented parents were asked if they gave their permission for the clinic to access their child's medical charts for use in the study. Parents were provided with HIPAA information sheets and an authorization form for release of their child's protected health information.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Parent of at least 1 child 6 months to 5 years old
* English-speaking or Spanish-speaking

Exclusion Criteria:

• N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2018-08-06 (Actual); Primary Completion 2019-03-28 (Actual); Study Completion 2019-11-25 (Actual)

PRIMARY OUTCOMES:
3-Month Change in Language Development | Baseline at enrollment to 3 months after enrollment
  3-month change in the percentage of child participants who achieved all age-appropriate language development milestones
3-Month Change in Social Development | Baseline at enrollment to 3 months after enrollment
  3-month change in the percentage of child participants who achieved all age-appropriate social development milestones
3-Month Change in Fine Motor Development | Baseline at enrollment to 3 months after enrollment
  3-month change in the percentage of child participants who achieved all age-appropriate fine motor development milestones
3-Month Change in Gross Motor Development | Baseline at enrollment to 3 months after enrollment
  3-month change in the percentage of child participants who achieved all age-appropriate gross motor development milestones

SECONDARY OUTCOMES:
3-Month Change in Family-Provider Communication | Baseline at enrollment to 3 months after enrollment
  3-month change in perception of the quality of communication between the family and provider
3-Month Change in Family-Provider Cultural Understanding | Baseline at enrollment to 3 months after enrollment
  3-month change in perception of the level of cultural understanding between the family and provider
3-Month Change in Family-Provider Cultural Concordance | Baseline at enrollment to 3 months after enrollment
  3-month change in perception of the importance of cultural concordance between the family and provider
Up-to-date Status of Well Child Visits | 12 months after study enrollment
  Up-to-date status of well child visits at 12 months
Up-to-date Status of Vaccination | 12 months after study enrollment
  Up-to-date status of vaccination at 12 months
Emergency Department Visits for Ambulatory-Sensitive Conditions | 12-month time period from study enrollment to 12 months after enrollment
  Number of emergency department visits for ambulatory-sensitive conditions from study enrollment to 12 months after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Ashaunta T Anderson, MD, MPH, Principal Investigator — Children's Hospital Los Angeles
Locations (1):
- Children's Hospital Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No